CLINICAL TRIAL: NCT02190669
Title: Exercise and Diabetes - an Observational Study of Exercise and Blood Glucose Control
Status: Completed | Type: Observational
Sponsor: Sansum Diabetes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 08-67
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- exercise in individuals without diabetes: exercise in individuals without diabetes
  Interventions: Other: exercise
- exercise in type 1 diabetes: exercise in type 1 diabetes
  Interventions: Other: exercise
- exercise in type 2 diabetes: exercise in type 2 diabetes
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Sprinting, walking on a treadmill, and stationary bicycle riding

SUMMARY:
This proposal seeks to gather continuous blood glucose and physical activity data from individuals with and without diabetes.

DETAILED DESCRIPTION:
This proposal seeks to gather continuous blood glucose and physical activity data from individuals with and without diabetes who are physically active and exercising for health benefits. The investigators hypothesize that insulin requirements will be inversely related to intensity of activity and an algorithm will be able to detect physical activity and automatically adjust insulin doses. Once such an algorithm has been determined for an individual, it can be applied to future similar situations, but ideally the algorithm will be dynamically refined based on closed-loop feedback information.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for subjects with diabetes
* Type 1 diabetes or insulin requiring type 2 diabetes for at least 1 year
* Use insulin to control diabetes
* Physically active (regularly work out, swim, run, walk, bike, etc.)
* Free of major micro- and macrovascular complications of diabetes
* 18-75 years of age
* A1C < 9.0% Inclusion criteria for subjects without diabetes
* No evidence of diabetes and physically active

Exclusion Criteria:

* unwilling to perform repeated glucose checks or take insulin as instructed
* abnormal thyroid function, kidney function, liver function
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals without diabetes and those with type 1 and type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Document the glycemic response of individuals without diabetes and with type 1 or type 2 diabetes | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Castorino, D.O., Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States